CLINICAL TRIAL: NCT05860946
Title: Safety and Efficacy of Remote Ischemic Conditioning in Adult Moyamoya Disease Patients Undergoing Revascularization Surgery
Brief Title: Remote Ischemic Conditioning in Adult Moyamoya Disease Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Heng Yang, Department of neurosurgery, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS9126
Record Dates: First submitted 2023-05-06; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Moyamoya Disease; Remote Ischemic Conditioning
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): Patients in RIC group and control group will achieve RIC intervention and sham RIC intervention three times daily from 5 days before operation and 7 days post operation
  Interventions: Device: Remote ischemic conditioning
- Control group (Sham Comparator): Patients in control group, bilateral upper arm cuffs were inflated to a pressure of 60 mm Hg for 5 minutes, followed by 5 minutes of relaxation of the cuffs
  Interventions: Device: Remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — The RIC intervention included five cycles of 5 min inflating tourniquets with the pressure of 200 mmHg and 5 min deflating with pressure of 0 mmHg alternately

SUMMARY:
Remote ischemic conditioning (RIC) is a non-invasive therapeutic approach for protecting organs or tissue against the detrimental effects of acute ischemia-reperfusion injury. Many protective factors produced by the stimulus of RIC could protect remote target organs and tissues through inhibiting oxidation and inflammation. The phenomenon of this protect effect was first found in myocardium ischemia-reperfusion injury and then RIC was used in children cardiac surgery to provide myocardial protection during operation. Then RIC was gradually applied to brain protection and a series of clinical researches have confirmed that it could improve the cerebral perfusion status, increase cerebral tolerance to ischemic injury, reduce perihematomal edema and promote clearance. Recently, a randomized controlled study reported that daily RIC could improve cerebral perfusion and slow arterial progression of adult MMD. Meanwhile, a single-arm open-label study also indicated that RIC was a promising noninvasive method for ischemic MMD control by relieving symptoms and reducing stroke recurrence. In addition, the effects of RIC on reducing neurological complications in MMD patients treated with revascularization surgery has also been reported. However, the mechanism of RIC in reducing peri-operative complications for MMD patients is still unknown. Thus, we conducted a randomized controlled study to explore the safety and efficacy of RIC in adult MMD patients undergoing revascularization therapy

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged from 18 to 65 years old;
2. Subjects all performed digital subtraction angiography (DSA) and diagnosed with MMD accroding to the criteria recommended by the Research Committee on MMD (Spontaneous Occlusion of the Circle of Wills) of the Ministry of Health and Welfare of Japan in 201211.
3. Modified Rankin Scale (mRS) score<4;
4. Informed consent obtained from the patient or legally authorized representative.

Exclusion Criteria:

1. Subjects suffered from acute ischemic or hemorrhagic stroke within 3 months;
2. Severe hepatic or renal dysfunction;
3. Severe cardiac disease;
4. Severe hemostatic disorder or severe coagulation dysfunction;
5. Serious, advanced, or terminal illnesses with anticipated life expectancy of less than one year;
6. Patients with moyamoya syndrome caused by autoimmune disease, Down syndrome, neurofibromatosis, leptospiral infection, or previous skull-base radiation therapy;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of major neurologic complications during perioperative period | 2 weeks after operation

SECONDARY OUTCOMES:
The Modified Rankin Scale (MRS) score | at 90 days postoperation and at 1 year after operation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang H, Hu Z, Gao X, Su J, Jiang H, Yang S, Zhang Q, Ni W, Gu Y. Safety and efficacy of remote ischemic conditioning in adult moyamoya disease patients undergoing revascularization surgery: a pilot study. Front Neurol. 2023 Jul 28;14:1200534. doi: 10.3389/fneur.2023.1200534. eCollection 2023. PMID 37576009